CLINICAL TRIAL: NCT01511081
Title: Randomized Phase II Study Comparing Stereotactic Body Radiotherapy (SBRT) With Stereotactic Body Proton Therapy (SBPT) for Centrally Located Stage I, Selected Stage II and Recurrent Non-Small Cell Lung Cancer
Brief Title: Stereotactic Body Radiotherapy (SBRT) Versus Stereotactic Body Proton Therapy (SBPT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-0691; P01CA021239 (NIH); NCI-2012-00071 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-10

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Non-small-cell lung cancer; NSCLC; Centrally-located; Recurrent; Squamous cell carcinoma; Adenocarcinoma; Large cell carcinoma; Bronchioloalveolar cell carcinoma; Non-small cell carcinoma not otherwise specified; Stereotactic Body Radiotherapy; SBRT; Stereotactic Body Proton Therapy; SBPT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Large Cell | interventions — Radiosurgery; Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBRT (stereotactic body radiotherapy) (Experimental): 50 Gy (RBE) in 4 daily treatments of stereotactic body radiotherapy (SBRT). Each treatment taking about 30-45 minutes per day.
  Interventions: Radiation: SBRT (stereotactic body radiotherapy)
- SBPT (stereotactic body proton therapy) (Experimental): 50 Gy (RBE) in 4 daily treatments of stereotactic body proton therapy (SBPT). Each treatment taking about 30-45 minutes per day.
  Interventions: Radiation: SBPT (stereotactic body proton therapy)

INTERVENTIONS:
Radiation: SBRT (stereotactic body radiotherapy) — 50 Gy (RBE) in 4 daily treatments of stereotactic body radiotherapy (SBRT). Each treatment taking about 30-45 minutes per day.
  Other Names: Radiotherapy; XRT
  Arms: SBRT (stereotactic body radiotherapy)
Radiation: SBPT (stereotactic body proton therapy) — 50 Gy (RBE) in 4 daily treatments of stereotactic body proton therapy (SBPT). Each treatment taking about 30-45 minutes per day.
  Other Names: Radiotherapy; XRT
  Arms: SBPT (stereotactic body proton therapy)

SUMMARY:
The goal of this clinical research study is to compare 2 types of radiotherapy, stereotactic body photon radiotherapy (SBRT) and stereotactic body proton radiotherapy (SBPT). Researchers would like to compare the side effects, quality of life, and cancer control.

DETAILED DESCRIPTION:
SBRT and SBPT:

Both SBRT and SBPT affect tumor cells in the same way. SBRT is the more common radiation technique of the two being studied and has been shown to be effective. However, SBRT may cause side effects when the tumor is close to normal organs because the photon does not stop totally after it hits the tumor cells.

SBPT is a type of radiation that uses charged-up particles. This beam of particles can be targeted like a laser to hit a tumor. When the beam travels through tissue, it starts to slow down. Doctors can control how deep the radiation particles go, to make sure that enough radiation hits the tumor being targeted and avoids the surrounding normal organs.

Both forms of radiation will be planned by a radiologist (radiation doctor) who will decide the dosage of radiation and how it will be given. Radiation technicians will follow the doctor's instructions to deliver your doses of radiation. Because your body moves during radiation, both photon and proton beams sometimes may have trouble staying on target. Proton radiation is more affected by the motion of your body than photon radiation. However, your doctors will use many methods to reduce motion.

Study Groups/Therapy:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in a flip of the coin) to 1 of 2 groups. You will have an equal chance of being in either group.

* If you are in Group 1, you will receive SBRT.
* If you are in Group 2, you will receive SBPT.

You will receive 4 treatments of SBRT or SBPT. During the treatment, you will lie still on a table for about 30-45 minutes per day in the same position for 4 days in a row.

You will not feel, see, or smell anything during the photon or proton beam delivery.

If you are randomly assigned to SBPT, a member of the radiation therapy staff will place 1-5 tiny metal pellets (called fiducial markers) around the tumor to help the radiation doctor locate the tumor during the daily proton therapy. The procedure could be done by a bronchoscopy or using a CT-guided needle placement through the chest wall.

Study Visits:

Once a week during the treatment:

* You will be asked about any side effects you may have had.
* You will have a physical exam.
* Your medical history will be recorded.

Length of Study:

You will finish study treatment after the 4th treatment of SBRT or SBPT. You will no longer be able to continue the same SBRT or SBPT to the same lesion if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions during the procedures. However, you can still receive other alternative treatments.

Follow-up Visits:

After the treatment, at 6 weeks, every 3 months (+/-1 month) for 2 years, every 6 months (+/-1 month) for 3 years, and then once a year for the rest of your life you will have follow-up. This follow-up schedule is standard of care.

* You will have a physical exam.
* Your medical history will be recorded.
* You will have a chest CT or PET scan to check the status of the disease.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Between 6 weeks and 6 months after treatment and then 1 time a year for 2 years, you will have a lung function tests.

On the 3rd or 4th follow-up visit and then 1 time a year for 2 years, you will have an ECG. A SPECT scan may be performed on the 3rd or 4th visit if the doctor thinks it is needed.

Your participation on the study will be over once you have completed the follow-up visits for 2 years. After the 2 years follow up, you will be followed according to the standard of care as described above. If the follow-up is at another hospital, the information about your medical history, physical exam, lung function, PET or CT scans will be sent to MD Anderson for review.

This is an investigational study. SBRT and SBPT are FDA approved for the treatment of lung cancer.

Up to 100 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation (by biopsy or cytology) or clinically diagnosed primary non-small cell lung cancer (NSCLC). The following primary cancer types are eligible: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, bronchioloalveolar cell carcinoma, or non-small cell carcinoma not otherwise specified
2. Centrally located, defined as located within 2 cm of the central bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, bronchus intermedius, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi), major vessels (aorta, pulmonary artery trunk, left/right pulmonary artery/vein main branches, superior/inferior vena cava, brachiocephalic artery trunk or left/right brachiocephalic vein, left/right subclavian artery/vein), esophagus, heart, tracheal, pericardium, mediastinal pleural and brachial plexus, chest wall and vertebral body, but no direct invasion, Stage I (T1-T2a <= 5 cm without main bronchus involvement), selective stage II ( selective T3 with involvement of mediastinal pleura, parietal pericardium,) based upon the following minimum diagnostic workup:
3. continued from criteria #2) History/physical examination including weight and assessment of Zubrod performance status within 2 months prior to registration; Evaluation by an experienced thoracic cancer clinician within 2 months prior to registration; computed tomography (CT) scan with intravenous contrast (unless medically contraindicated) of the entirety of both lungs and the mediastinum, most part of liver, and adrenal glands acquired within 2 months prior to registration must be available. The primary tumor dimension will be measured on the CT in lung window. If PET/CT is performed within 2 month prior to registration, CT of chest is recommended but nor required. Whole body fluorodeoxyglucose positron emission tomography (FDG-PET) within 3 months prior to registration with adequate visualization of the primary tumor and draining lymph node basins in the hilar and mediastinal regions and adrenal glands; Pulmonary function tests (PFTs):
4. continued from inclusion #3) Routine spirometry, lung volumes, diffusion capacity (within 3 months prior to registration). Patients with hilar or mediastinal lymph nodes </= 1cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may still be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer. The primary tumor should be considered medically inoperable by an experienced thoracic cancer clinician for a standard lobectomy and mediastinal lymph node dissection/sampling procedure or patient refuses surgery. The patient may have underlying physiological medical problems that would prohibit a surgery due to a low probability of tolerating general anesthesia, the operation, the postoperative recovery period, or the removal of adjacent functioning lung.
5. continued from inclusion #4) These types of patients with severe underlying health problems are deemed "medically inoperable." Standard justification for deeming a patient medically inoperable based on pulmonary function for surgical resection of NSCLC may include any of the following: Baseline forced expiratory volume in 1 second (FEV1) < 50% predicted, postoperative FEV1 < 30% predicted, severely reduced diffusion capacity, baseline hypoxemia and/or hypercapnia, exercise oxygen consumption < 50% predicted, severe pulmonary hypertension, diabetes mellitus with severe end organ damage, severe cerebral, cardiac, or peripheral vascular disease, or severe chronic heart disease. If the patient has medically resectable/operable disease but declines surgery after consulting with a thoracic surgeon, he/she will be considered eligible.
6. History of NSCLC treated with surgery and/or radiotherapy previously and disease has been cured or clinically no disease progression for more than 6 months, now isolated recurrent disease in lung parenchyma and without involvement of main bronchus, chest wall, hilar/mediastinal lymph nodes and critical mediastinal structures. Biopsy of recurrent disease is recommended.
7. Zubrod Performance Status 0-2;
8. Age >/= 18
9. Women of childbearing potential and male participants must agree to use a medically effective means of birth control, such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills, throughout their participation in the treatment phase of the study.
10. The patient must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Direct evidence of hilar or mediastinal lymph nodes or distant metastases after appropriate staging studies.
2. Patients with active pulmonary or pericardial infection.
3. Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
4. Patient pulmonary function showed that pre-bronchial dilator FEV1 <25% or DLCO<25%.
5. Patient currently requiring supplemental oxygen for his/her daily life.
6. Patient is pacemaker dependent.
7. Patients </= 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Y. Chang, MD, MS, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 28, 2012 to August 31, 2015. Recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 21 participants enrolled, four were excluded from the study before assignment to groups.
Period: Overall Study
Arm/Group | SBRT (Stereotactic Body Radiotherapy) | SBPT (Stereotactic Body Proton Therapy)
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBRT (Stereotactic Body Radiotherapy) | SBPT (Stereotactic Body Proton Therapy) | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Median (Full Range); unit: years] | 77 [66 to 88] | 72 [57 to 87] | 74 [57 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Summary of 2-Year Stereotactic Body Radiotherapy (SBRT) and Stereotactic Body Proton Therapy (SBPT) Related Toxicities by Grade 3+ Treatment-related Toxicity
Description: Outcome defined as 2-year rate of stereotactic body radiotherapy (SBRT)- and SBPT-related toxicities according to Common Terminology Criteria for Adverse Events (CTCAE) v.4 criteria, including: radiation-induced pneumonitis/fibrosis/fistula, esophagitis/stricture/fistula.
Time Frame: 2 years
Population: Early study termination. Inadequate enrollment and study period to complete analysis per protocol.
Arm/Group | SBRT (Stereotactic Body Radiotherapy) | SBPT (Stereotactic Body Proton Therapy)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Treatment Response
Description: Prospective assessment of positron emission tomography (PET) standardized uptake value (SUV) changes as a measure of treatment response and outcomes. Pulmonary function changes as a function of treatment and response.
Time Frame: 2 years
Population: Early study termination. Inadequate enrollment and study period to complete analysis per protocol.
Arm/Group | SBRT (Stereotactic Body Radiotherapy) | SBPT (Stereotactic Body Proton Therapy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be evaluated weekly during the course of treatment, four treatments of SBRT or SBPT expected.
Arm/Group | SBRT (Stereotactic Body Radiotherapy) | SBPT (Stereotactic Body Proton Therapy)
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT (Stereotactic Body Radiotherapy) (N=8) | SBPT (Stereotactic Body Proton Therapy) (N=9)
Metastatic squamous cell carcinoma of the lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects to be analyzed none meeting the two year reporting period for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes